CLINICAL TRIAL: NCT03540095
Title: Randomized Prospective Clinical Trial of Erector Spinae Plane (ESP) Versus Paravertebral Nerve (PVB) Blockade for Acute Unilateral Rib Fracture Pain
Brief Title: Erector Spinae Plane (ESP) Versus Paravertebral Nerve (PVB) Blockade for Acute Unilateral Rib Fracture Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to staffing issues, we are unable to enroll patients at the clinical site assigned. The study is terminated.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Samuel Goldstein, Anesthesia Resident, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO18040578
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Rib Fractures; Pain, Acute; Thoracic Injuries; Neuropathic Pain; Neuromuscular Blockade; Anesthesia, Local
MeSH Terms: conditions — Rib Fractures; Acute Pain; Thoracic Injuries; Neuralgia

STUDY DESIGN:
Intervention Model Description: There are two arms. Our 60 patients will be randomized to either of the two arms and studied in parallel.
Masking Description: We are unable to mask the patient or provider for this study. The interventions are inherently similar, but different, thus making it impossible to blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Experimental): The patients randomized to the Erector Spinae Plane Block arm will receive this nerve block at the level corresponding to the rib fractures. Ropivicaine 0.5% 25 mL will be used during the procedure for initiation of pain control. Bupivicaine 0.0625% will be used for continuous infusion of local anesthetic. It will be titrated to effect, at maximum 12 mL/hr. Bupivicaine 0.0625% 3mL will be given every hour as a bolus additionally.
  Interventions: Drug: Erector Spinae Plane Block
- Paravertebral Nerve Block (Experimental): The patients randomized to the Paravertebral Nerve Block arm will receive this nerve block at the level corresponding to the rib fractures. Ropivicaine 0.5% 25 mL will be used during the procedure for initiation of pain control. Bupivicaine 0.0625% will be used for continuous infusion of local anesthetic. It will be titrated to effect, at maximum 12 mL/hr. Bupivicaine 0.0625% 3mL will be given every hour as a bolus additionally.
  Interventions: Drug: Paravertebral Nerve Block

INTERVENTIONS:
Drug: Erector Spinae Plane Block — See arm description
  Other Names: Ropivicaine 0.5%; Bupivicaine 0.0625%; Braun 18 Ga x 3.5 in TUOHY Epidural Needle; Braun 20 Ga CLOSED TIP CATHETER; Sonosite X-Porte portable ultrasound machine
  Arms: Erector Spinae Plane Block
Drug: Paravertebral Nerve Block — See arm description
  Other Names: Ropivicaine 0.5%; Bupivicaine 0.0625%; Braun 18 Ga x 3.5 in TUOHY Epidural Needle; Braun 20 Ga CLOSED TIP CATHETER; Sonosite X-Porte portable ultrasound machine
  Arms: Paravertebral Nerve Block

SUMMARY:
Continuous paravertebral analgesia and erector spinae plane blockade (ESP) are accepted techniques at University of Pittsburgh Medical Center (UPMC) for the management of thoracic pain following surgery and trauma. Recently, an increasing number of erector spinae plane blocks are being performed as it has been demonstrated in our institution and via case reports that they provide clinical effectiveness, but may have a better side-effect profile than the paravertebral nerve block. However, the relative efficacy of ESP and continuous paravertebral analgesia for patients with rib fractures remains to be established. This study will include 60 consecutive patients presenting to the UPMC Presbyterian Acute Interventional Perioperative Pain Service suffering from unilateral rib fractures and will be randomized to receive either nerve blocks via continuous paravertebral infusion or via erector spinae plane infusion. In addition, to treat breakthrough pain, the patients in both arms will receive multimodal adjunctive therapy per routine. Bupivicaine and ropivicaine are FDA approved for use in nerve block catheters. The primary outcome will be total opioid consumption in the first 3 days of nerve block. Secondary outcomes include highest visual analog pain score (VAS) with deep breathing and at rest, adverse events, and total number of nerve blocks. Other data points include time to readiness for discharge, and length of hospital stay.

DETAILED DESCRIPTION:
All interventions regarding the placement and management of ESP and paravertebral blocks in this study are consistent with existing standard of care practices at UPMC and utilize protocols that are already in use. In addition, by nature of being included in a research study, patients are likely to receive closer monitoring for side-effects.

Screening and enrollment: After approval by the institutional review board, all (American Society of Anesthesiology) ASA I-IV patients aged 18-85 years, weighing between 50 and 120 kg with unilateral rib fractures will be screened for enrollment. Sixty patients will be enrolled in this randomized prospective study with equal numbers in each arm of the trial. This study design is unblinded as we cannot blind patients nor observers as to the type of block performed (slightly different location). This is an accepted limitation of the study. No advertising will be used and no monetary compensation will be offered. The nature of the study, planned interventions, risks, benefits, and alternatives will be discussed in detail with the patients at the time of enrollment and prior to the patients' signing of a written consent form.

Randomization: Patients will be enrolled into one of the study groups on the day of consultation in an alternating fashion. The study groups are defined as: Group I: Erector Spinae Plane Block (ESP) 30 patients Group II: Paravertebral Block (PVB) 30 patients.

Day of Block: After written informed consent is confirmed, a research assistant will introduce the scoring system used for pain assessment (VAS), and demonstrate proper use of the incentive spirometer.

All nerve blocks will be performed by an experienced member of UPMC's pain management service. Both nerve blocks can take between 10-60 minutes to perform. They will either occur in the ICU or on a monitored medicine floor.

Paravertebral nerve block catheter placement and activation (PVB group only): Paravertebral catheters will be placed according to UPMC standard of care practices as outlined below: After an intravenous catheter has been established and standard monitors and oxygen applied, the patient will be placed in the sitting position. The patient will be administered appropriate sedation based on the discretion of the provider if needed to safely perform the procedure.

Paravertebral technique: With the patient in a sitting position, the point of needle entry will be marked on the skin corresponding to paravertebral catheter placement. The thoracic spine level will be at the anatomic level corresponding to the ribs fractured. The needle entry sites will be 2.5 cm lateral to the midpoint of the spinous process of the corresponding thoracic vertebrae. The area will be prepped and draped in a sterile fashion, and 1% lidocaine infiltrated subcutaneously at each point of anticipated needle entry. For each of the catheter placement, a sterile gauge Tuohy needle will be introduced with ultrasound guidance towards the paravertebral space. After final needle placement, a hanging drop technique will be used to assess for interpleural placement while the patient inhales and exhales deeply. Next 5 mL of ropivicaine 0.5% will be injected incrementally through each needle after negative aspiration under ultrasound visualization, followed by insertion of the nerve block catheter to a depth 5 cm beyond the tip of the needle. An additional 20 mL of ropivicaine 0.5% will then be injected in 5 mL increments with negative aspiration in between, through each catheter yielding a total activation dose of 25 ml of ropivicaine 0.5% via each catheter. The catheters will be secured with Steri-strips and a transparent occlusive dressing. Vital signs will be monitored at regular intervals until the procedure is complete.

Erector spinae catheter placement and activation (ESP group only): An erector spinae plane catheter will be placed according UPMC standard of care practices as outlined below: After an intravenous infusion has been established and standard monitors and oxygen applied, the patient will be placed in the sitting position. The patient will be administered appropriate sedation based on the discretion of the provider if needed to safely perform the procedure.

ESP technique: With the patient in a sitting position, the point of needle entry will be marked on the skin corresponding to the appropriate vertebral level relative to the rib fractures. The area will be prepared and draped in a sterile fashion, and 1% lidocaine infiltrated subcutaneously at the point of anticipated needle entry. A sterile Tuohy needle will be introduced and advanced towards the corresponding transverse process. Hydrodissection will ensure that the proper plane is located. Once the erector spinae musculature is separated from the rib, 25ml of ropivicaine 0.5% will be introduced into the plane under ultrasound guidance. A catheter will be placed to a depth 5 cm beyond the tip of the needle. The catheter will be secured with Steri-strips and a transparent occlusive dressing. Vital signs will be monitored at regular intervals until the procedure is completed.

Paravertebral infusions of Bupivicaine 0.0625% will be titrated to 12 ml/hr maximum for the patients in the paravertebral catheter group (Group PVB). Patients in the ESP group (ESP) will start a continuous infusion of Bupivicaine 0.0625% and titrate to 12 mL/hr maximum as needed for pain. The patients in both groups will also be given access to acetaminophen 1000 mg every 6 hours IV or PO if there is no contraindication. Other adjuncts such as gabapentin, celebrex, ketamine, and opioid analgesics may be adjusted by the physicians involved based on the patients clinical condition. A PCA may be required for opioid pain medication administration initially, and will be continued until the patient is able to tolerate oral pain medication. Additional pain relief is available via nurse-administered 3 mL boluses of 0.0625% bupivacaine via the catheter pumps.

Post nerve block anesthesia protocol: Once on the floors, additional pain relief is available via nurse-administered 3 mL boluses of Bupivicaine via the catheter pumps given no more than hourly. All patients will be assessed daily by members of the acute interventional perioperative pain service. The infusion rates via the paravertebral and ESP catheters may be adjusted at the discretion of the pain service up to a rate of 12 mL/hr on each side (standard infusion rate used at UPMC-Presbyterian). All paravertebral ESP catheters will be stopped and removed as tolerated by the patient or post-procedure day #5, whichever occurs first. Additional pain medication will be available to all patients per standard of care.

ICU (Intensive Care Unit): Patients will be admitted to an intensive care unit at the discretion of the emergency department. Patients who are intubated and sedated, and who are unable to participate medical decision making will not be accepted for this study. If a patient fits the inclusion criteria and is in the ICU, the nerve block will be placed and managed in the ICU as above for all other situations.

Data will be collected daily from the patients until the nerve block is removed or 5 days post-procedure, whichever comes first.

Discharge: The readiness for discharge will be determined by the primary team: This decision will likely include (1) return of respiratory function, (2) hemodynamic stability, (3) normothermia, (4) no clinical evidence of DVT/PE (Deep Vein Thrombosis/Pulmonary Embolism) which is untreated, (5) pain controlled by oral agents. In addition, actual length of hospital stay will be recorded. Nerve block will be performed and the catheters will be removed according to the ASRA (American Society of Regional Anesthesia and Pain Medicine) guidelines for regional anesthesia catheter placement and removal available on the ASRA website.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-85 years
* no contraindications to the placement of a paravertebral catheter or erector spinae plane catheter
* American Society of Anesthesiologists physical status between I-IV
* no chronic opioid use
* patients who are not expected to be on therapeutic anticoagulants post-procedurally
* no clopidogrel in last 48 hours
* no known allergies to any of the drugs/agents used study protocol
* no personal or family history of malignant hyperthermia
* not pregnant
* not having an altered mental status (oriented to place, person, or time)
* no comorbid condition(s) that in the judgment of the anesthesiologist, would preclude the patient from any aspect of the study. Comorbid conditions include bleeding disorders, thrombocytopenia, localized infection, sepsis, possibly abnormalities of the thoracic spine or paravertebral anatomy neoplastic mass occupying the paravertebral space, empyema, allergy to local anesthestic drug, increased intracranial pressure, severe uncorrected hypovolemia, fixed cardiac output states.

Exclusion Criteria:

* Age younger than 18 years or older than 85 years
* any contraindication to the placement of a paravertebral or erector spinae catheters
* American Society of Anesthesiologists physical status V or greater
* chronic opioid use
* coagulation abnormalities or patients who are expected to be on therapeutic anticoagulants postprocedurally
* clopidogrel use within 48 hours
* allergy to any of the drugs/agents used study protocol
* personal or family history of malignant hyperthermia
* pregnancy
* having an altered mental status (not oriented to place, person, or time), (11) any comorbid condition that in the judgment of the anesthesiologist would preclude the patient from any aspect of the study
* patient refusal. Comorbid conditions include bleeding disorders, thrombocytopenia, localized infection, sepsis, possibly abnormalities of the thoracic spine or paravertebral anatomy neoplastic mass occupying the paravertebral space, empyema, allergy to local anesthetic drug, increased intracranial pressure, severe uncorrected hypovolemia, fixed cardiac output states.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Total Opioid Consumption | first 72 hours after intervention

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Pain Scores | Immediately prior to intervention. 15 minutes after intervention. 60 minutes after intervention. Daily (in morning) for 3 total days after intervention.
  Visual Analog Scale is numerical from 0-10, with 10 being the worst pain imaginable, and 0 being no pain. The pain score will be recorded at rest and with deep breathing at the time intervals below. There are no subscales involved in this measurement. Simply, we will record single pain scores by VAS scale at rest and with deep breathing at indicated times.
Adverse Events | During the expected duration of this study, which is on average 5 days.
  We will record total number of pneumothoraxes, site infections, significant bleeding events, and unintentional catheter removals. Each of these events will be added separately per patient. We will analyze how many patients experience any adverse effect, and then further study the incidence of each specific adverse effect and compare them across both interventions.
Number of Nerve Blocks | During the expected duration of this study, which is on average 5 days.
  The provider will use his/her judgement to determine how many nerve blocks are required for management of the rib fracture pain. Compare the number of nerve blocks required for each type of intervention in the separate arms.
Length of Stay | Will evaluate length of stay upon termination of the last study subject. Expected to be within 6 months of initiation of the trial.
  Total length of hospitalization
Time until discharge | Will evaluate length of stay upon termination of the last study subject. Expected to be within 6 months of initiation of the trial.
  Time from intervention to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Goldstein, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center - Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No